CLINICAL TRIAL: NCT00491790
Title: Montelukast With Status Asthmaticus, Ages 2-5
Status: Unknown | Phase: Phase 2 / Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD) (NIH)
Collaborators: Pediatric Pharmacology Research Units Network (Network)
Responsible Party: Jeffrey L. Blumer, Ph.D, M.D., University Hospitals Case Medical Center
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: PPRU 10854
Record Dates: First submitted 2007-06-22; First posted 2007-06-26 (Estimated); Last update posted 2008-12-16 (Estimated); Status verified 2008-11

CONDITIONS: Status Asthmaticus; Asthma
Keywords: montelukast; Albuterol; Status Asthmaticus; Asthma
MeSH Terms: conditions — Status Asthmaticus; Asthma | interventions — montelukast

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1 (Sham Comparator): Sterile Water
  Interventions: Other: Sterile water
- Montelukast (Active Comparator): Dissolved granules in sterile water
  Interventions: Drug: Montelukast

INTERVENTIONS:
Drug: Montelukast — Montelukast 4 mg rapid dissolving granules in sterile water given orally once
  Arms: Montelukast
Other: Sterile water — Sterile water
  Arms: 1

SUMMARY:
The purpose of this study is to determine if montelukast, in addition to standard treatment is helpful in treating patients ages 2-5 who are in the hospital because of status asthmaticus.

DETAILED DESCRIPTION:
This is a prospective study of montelukast efficacy in addition to standard treatment of status asthmaticus in children from 2-5 years old who are in the PICU. Children who meet eligibility requirements will be randomized to receive a rapid-dissolving oral dose of montelukast or placebo. Once enrolled, a baseline modified Wood's-Downes clinical asthma severity score will be recorded pre and post completion of a standard nebulized albuterol treatment of 0.15 mg/kg/dose (min2.5mg/dose). Patients who are able will have FEV1 measurements obtained at predetermined intervals for determination of clinical asthma severity score. Blood samples for PK analysis will be collected prior to study drug administration and at predetermined time intervals to determine the plasma level of montelukast. In addition, a blood sample will be obtained for genetic study of polymorphisms of CYP3A4, CYP3A5, and CYP2C9.

ELIGIBILITY:
Inclusion Criteria:

* Participant's parent/legal guardian must give written informed consent prior to study participation. When appropriate, written assent from the child will also be obtained.
* Participant, male or female, must be 2 to 5 years of age.
* Participant must have a history of reactive airway disease (RAD) or asthma, and must currently be admitted for an acute exacerbation of RAD or asthma.
* Primary physician must believe that patient would benefit from improved bronchodilation and improvement in clinical asthma severity score.
* Participant must have received standard therapy for status asthmaticus: Oxygen as needed; 3 nebulized albuterol treatments of at least 2.5mg/dose; Methylprednisolone or prednisone loading dose of 2mg/kg; Ongoing methylprednisolone therapy @ 0.5mg/kg every 6

Exclusion Criteria:

* Known hypersensitivity to montelukast
* Chronic lung disease
* Cardiac or pulmonary congenital anomalies
* Known renal disease
* Known hepatic disease
* Known immunologic disorders other than allergy and atopy
* Other explanations for respiratory distress
* Use of leukotriene modifiers within 2 weeks of the acute presentation
* Intubated patients

Ages: 2 Years to 5 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 52 (Estimated)
Dates: Start 2006-12; Primary Completion 2010-01 (Estimated); Study Completion 2010-10 (Estimated)

PRIMARY OUTCOMES:
Effectiveness of Montelukast as adjunctive therapy

SECONDARY OUTCOMES:
Estimate the first dose pharmacokinetic parameters of Montelukast

CONTACTS AND LOCATIONS:
Overall Officials: Jeffrey L. Blumer, M.D., Ph.D., Principal Investigator — PPRU
Locations (1):
- Rainbow Babies and Children's Hospital, Cleveland, Ohio, United States